CLINICAL TRIAL: NCT07261371
Title: A PHASE 1, OPEN LABEL, SINGLE DOSE, RANDOMIZED, CROSSOVER STUDY TO EVALUATE THE BIOEQUIVALENCE OF TWO FORMULATIONS OF A CGRP RECEPTOR ANTAGONIST IN HEALTHY ADULT PARTICIPANTS
Brief Title: A Study to Compare Blood Levels of Two Different Dosage Formulations of the Study Medicine Called CGRP Receptor Antagonist in Healthy Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: C4951081
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteer
Keywords: Healthy volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Sequence 1 (Experimental)
  Interventions: Drug: Test formulation (Treatment A); Drug: Reference formulation (Treatment B)
- Treatment Sequence 2 (Experimental)
  Interventions: Drug: Test formulation (Treatment A); Drug: Reference formulation (Treatment B)

INTERVENTIONS:
Drug: Test formulation (Treatment A) — calcitonin gene-related peptide receptor inhibitor
Drug: Reference formulation (Treatment B) — calcitonin gene-related peptide receptor inhibitor

SUMMARY:
The purpose of this study is to assess the bioequivalence (medicines that may have different names or be made in different ways, but have the same effect on the body) of different formulations of a CGRP receptor antagonist in healthy adult participants.

The study is seeking participants who are:

1. Healthy males and females 18 years of age or older
2. Willing and able to comply with all scheduled visits, treatment plan, lifestyle considerations, and other study procedures.
3. Body Mass Index of 16-32 kilogram per meter squared (kg/m2); and a total body weight >45 kg

The study will help the team understand how difference in formulation may, or may not, affect how the medicine is absorbed, processed, and removed by the body.

ELIGIBILITY:
Inclusion:

1. Male and/or female participants must be 18 years of age or older (or the minimum age of consent in accordance with local regulations) at screening who are overtly healthy as determined by medical evaluation including medical history, physical examination, and laboratory tests.
2. BMI of 16-32 kg/m2; and a total body weight >45 kg.
3. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.

Exclusion:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Any medical, psychiatric condition, suicidal ideation and behavior, laboratory abnormality or other conditions that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
3. Use of prescription or nonprescription drugs and dietary and herbal supplements within 14 days or 5 half lives (whichever is longer) prior to the first dose of study intervention.
4. Previous administration of an investigational product (drug or vaccine) within 30 days or 5 half lives preceding the first dose of study intervention used in this study (whichever is longer). Participation in studies of other investigational products (drug or vaccine) at any time during participation in this study.
5. A positive urine drug test. A single repeat for positive drug screen may be allowed.
6. Unwilling or unable to comply with the Lifestyle Considerations criteria of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2026-05-08 (Estimated); Study Completion 2026-05-08 (Estimated)

PRIMARY OUTCOMES:
Area under the Plasma Concentration-Time profile from time 0 extrapolated to infinite time (AUCinf) of the test and reference formulations | Pre-dose to 72 hours
Area under the Plasma Concentration-Time profile from time 0 to time of last quantifiable data point (AUClast) of the test and reference formulations | Pre-dose to 72 hours
Maximum Observed Plasma Concentration (Cmax) of test and reference formulations | Predose to 72 hours

SECONDARY OUTCOMES:
Number of participants with Clinically Significant Abnormalities in Laboratory Parameters | Baseline up to 36 days after the last dose of study intervention
Number of Participants with Treatment Emergent Adverse Events (TEAEs) | Baseline up to 36 days after the last dose of study intervention

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - New Haven, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4951081